CLINICAL TRIAL: NCT00184470
Title: Mapping of Traumatized Patients Referred to St. Olavs Hospital in the Period 2000-2003-Norwegian University of Science and Technology
Brief Title: Trauma Registration at St. Olavs Hospital 2000-2003
Status: Terminated | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Other Study IDs: NTNU-Traume-1
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Injuries, Multiple; Norway/Epidemiology; Trauma Centers/Statistics & Numerical Data; Trauma, Multiple; Trauma Severity Indices
Keywords: Adult; Child; Hospitalization/statistics & numerical data; Retrospective studies
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
St. Olavs Hospital is a trauma referral center in the region of Midtnorge. Admitting trauma patients locally and those referred from hospitals in Nord-Trøndelag, Sør-Trøndelag and Møre-Romsdal.An active trauma team was defined in 1992, but it's work has not been evaluated earlier. Prospective studies of these patients were established 1st of January 2004 at St. Olavs Hospital.

DETAILED DESCRIPTION:
This mapping is a observational retrospective study of trauma patients admitted to St.Olavs Hospital from 2000 until 2003. Patient journals (electronic and paper), autopsy reports and the emergency medical respons systems (AMK) database have been reviwed. We are reviewing the local traumaepidemiology, traumateam performance, mechanisms of injury and the potenially avoidable deaths in trauma.

ELIGIBILITY:
Inclusion Criteria:

* Trauma team activation
* Motor vehicle crash with ejection
* Pedal cyclist, motorcyclist or pedestrian hit by vehicle >30 km/h
* Fall > 5 meters
* Fatality in same vehicle
* Interhospital trauma transfer within 24 hrs
* Injury to two or more body regions
* Fracture to two or more long bones
* Spinal cord injury
* Amputation of a limb
* Penetrating injury to head, neck, torso or proximal limb

Exclusion Criteria:

* Burns
* Strangulations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Skogvoll, MD, PhD, Study Director — Norwegian University of Science and Technology